CLINICAL TRIAL: NCT01729221
Title: Application of the Stem Cell Therapy in the End Stage Liver Disease and Assessment Its Consequences in the Quality of Live Style as Well as Development of HCC.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zekri AR, Proffesor, Cairo University
Other Study IDs: 1
Record Dates: First submitted 2012-11-17; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Hepatocellular Carcinoma in Hepatitis C Virus Infected Patients
Keywords: Hepatocellular carcinoma; Hepatitis C virus
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HCV infected patients treated by stem cell therap: Hepatitis C virus infected patients treated by stem cell therapy
- HCV infected patients treated by standared line of care: Hepatitis C virus infected patients treated by standared line of care

SUMMARY:
Prospective study to calculated the incidence of hepatocellular carcinoma in hepatitis C virus infected patients after stem cell therapy.

DETAILED DESCRIPTION:
Our prospective research is carried out in one of the stem cell therapy centers in Egypt where 140 hepatitis C virus infected patients attending for stem cell therapy are enrolled in our study and the patients will be followed up after stem cell therapy where the incidence of hepatocellular carcinoma after stem cell therapy will be calculated , another group of hepatitis C virus infected patients attending to Kasr El Aini university hospital to receive the standered line of care as indicated will be enrolled in our study and will be followed up , where the incidence of hepatocellular carcinoma will be calculated and compared to the previous group , to determine if there is a significant difference between both groups regarding the incidence of hepatocellular and determine whether stem cell therapy affecets the incidence of hepatocellular carcinoma in hepatitis C virus infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged from 20 to 65 years of age.
* Evidence of chronic liver insufficiency.
* The presence of decreased serum albumin and/or increased bilirubin and/or increased international normalized ratio (INR).
* Patient is unlikely to receive a liver transplant.
* Ability to give written consent
* Women of childbearing potential may be included, but must use a reliable and appropriate contraceptive method

Exclusion Criteria:

* Patients below the age of 20 or above the age of 65 years
* Pregnant or lactating women
* Patients with recent recurrent GI bleeding or spontaneous bacterial peritonitis
* Patients with evidence of HIV or other life threatening infection
* Patients unable to give informed consent
* Patients with a history of hypersensitivity to G-CSF
* Patients who have been included in any other clinical trial within the previous month
* Patient with recurrent attacks of hepatic encephalopathy.
* Evedince of portal vein thrombosis by ultrasound.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis C virus infected patients indicated for stem cell therapy
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-02 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of hepatocellular carcinoma post stem cell therapy in hepatitis C virus infected patients | within the first year after stem cell therapy

SECONDARY OUTCOMES:
Compare the incidence of hepatocellular carcinoma in patients who had received stem cell therapy to those who had received the standared line of care | within one year of follow up of hepatitis C virus infected patients

OTHER OUTCOMES:
Compare liver function in both groups | after one year of follow up
asses liver functions in both groups | after one year of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Zekri Abdelrahman, M.SC, Ph,D, Study Chair — National Cancer Institute , Cairo University; Hosny Salama, M.D., Study Director — Cairo University; Zekri Abdelrahman, M.SC, Ph,D, Principal Investigator — National Cancer Institute, Cairo University
Locations (1):
- Cairo University & National Cancer Institute, Cairo, Egypt

REFERENCES:
- [Derived] Salama H, Zekri AR, Medhat E, Al Alim SA, Ahmed OS, Bahnassy AA, Lotfy MM, Ahmed R, Musa S. Peripheral vein infusion of autologous mesenchymal stem cells in Egyptian HCV-positive patients with end-stage liver disease. Stem Cell Res Ther. 2014 May 28;5(3):70. doi: 10.1186/scrt459. PMID 24886681